CLINICAL TRIAL: NCT03911830
Title: Effects of an Aerobic Exercise Program on Cycloergometer Followed by Cold Water Immersion Recovery in Patients With Rheumatoid Arthritis
Brief Title: Aerobic Exercise Program Followed by Cold Water Immersion: Effects on Arthritis Patients Arterial Stiffness
Acronym: PREXCRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P/2016/305
Record Dates: First submitted 2018-10-01; First posted 2019-04-11 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis; Cryotherapy Effect; Physical Activity
Keywords: Rheumatoid Arthritis; Physical exercise; Cryotherapy; Pulse Wave Velocity
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise followed cold water immersion (Experimental): Exercise program on cycloergometer and its submerged recovery
  Interventions: Other: Exercise followed cold water immersion

INTERVENTIONS:
Other: Exercise followed cold water immersion — Rehabilitation program of 17 sessions with 30 minutes of exercise followed by 15 minutes of submerged recovery at 17 ° C (3 sessions per week / 6 weeks).

SUMMARY:
The purpose of this study is to analyze the long-term effects of a physical exercise program on the cardiovascular system of people with Rheumatoid Arthritis (RA).

Indeed, it is recognized that RA patients have cardiovascular problems and that regular physical exercise (exercise training) may be beneficial for the disease complications, incluse the cardiovascular risk. Unfortunately, these patients do not exercise enough for fear of joint pain or for fear of deteriorating their general physical condition.

It is known that intermittent exercises, ie combining low and high intensity work phases, are particularly effective in the cardiovascular field. As it is possible that the high intensity phases be more difficult to sustain than the low intensity phases (joint pain and degradation of the inflammatory status), the investigators propose to study the effects of cold water immersion in the legs after performing this exercise, because the cold being recognized as limiting the pain and improving the inflammatory status.

DETAILED DESCRIPTION:
The first visit or selection visit, will be the opportunity for the investigator to submit the Information Notice and Informed Consent about. A second visit or visit of inclusion will be the occasion of the return of the signed informed consent of the subject. This visit will include a clinical examination for the detection of a pathology likely to contraindicate the practice of a physical activity and a resting electrocardiogram. The investigator will record the data for each subject, and check the eligibility criteria. Patient's treatments will not be interrupted throughout the program.

The typical rehabilitation sessions will be performed according to the intermittent exercise followed by a cold water immersion recovery at 17 ° Celsius for 15 minutes. The total duration of the rehabilitation session will be approximately 50 minutes and the sessions should be separated by at least 48 hours with a frequency of 3 sessions per week by 6 weeks, totalizing 17 sessions.

The typical sessions will be conducted as follows: intermittent exercise on a cycle ergometer for 30 minutes in sub-maximal intensity; application of the BORG scale; immersion in cold water at 17 ° C for 15 minutes and application of the cold water tolerance scale. The subject's heart rate will be recorded continuously for the duration of the sessions by a heart rate monitor (Polar Electro, Finland).

Intermittent exercise consists of six 5-minute cycles with a succession of work (high: 1 minute, moderate: 4 minutes). The high intensity work phase will be adjusted to achieve a target Heart Rate (HR) corresponding to HR rest + 70% HR reserve (HR reserve = (200 - age) - HR rest). The low intensity work phase will be adjusted to achieve a maximum target HR corresponding to HR rest + 50% HR reserve. In total, the exercise has a sub maximal intensity, commonly used in exercise rehabilitation studies conducted on various pathologies. It is an intensity capable of promoting cardiovascular benefits without representing a severe intensity for the patient.

The target intensity for intermittent work is controlled by monitoring the HR. To achieve the desired , patients will be asked to adjust their pedaling frequency. The patient therefore adapts his pedaling frequency in accordance with the target HR to switch from one workload to another. During the rehab sessions, the wattage and pedaling frequency will be recorded. The cycloergometer used will be of the brand Monark (type 839E).

Measurements will be made before, in the middle and at the end of the program (before 1st, 10th and after 17th session (S1, S10 & S17). These examinations are commonly performed in the follow-up of rheumatoid arthritis:

1. / The blood sample will be taken at the elbow crease by a clinical research nurse. There will be a total of three blood samples of approximately 7 mL of blood for subjects who are doing the entire program and only two blood tests for other subjects. Venous blood samples will be used to determine serum marker concentrations of C-reactive protein inflammation. The investigators will also perform the assay of two other blood markers of IL-6 inflammation and TNF-alpha classically used in the clinical follow-up of this kind of patient.
2. / The clinical examinations will consist in the evaluation of the DAS-28 as well as an ultrasound of the joints. The Disease Activity Score (DAS) and its derivatives have been developed and validated by Dutch authors and considered the best test for the RA classification by the European League Against Rheumatism (EULAR). Several studies have shown that there is a very good correlation between the evaluation of RA activity on only 28 joints compared to 44 or 66. DAS-28 includes pain rating for joint pressure and joint swelling on the proximal interphalangeal (PPI), metacarpophalangeal (MCP) joints of the hands, wrists, elbows, shoulders, and knees. DAS-28 has the advantage of being more quickly achieved and of not rating rare joints such as distal interphalangeal or temporomandibular. It is however often criticized because it does not evaluate the joints of the feet which are on the contrary very frequently painful or inflammatory in this disease. Nevertheless, DAS-28 is currently the most frequently used score for the assessment of RA activity, whether in clinical studies or in routine practice.

   The articular ultrasound will be performed with an ESAOTE mylab five device on 32 joints of the hands, wrists and feet using a qualitative synovitic score in B mode and Doppler mode, each rated from 0 to 32, for a total score ranging from 0 to 64.
3. / The assessment of functional disability, physical activity and quality of life and well-being will be done using questionnaires: HAQ, SQUASH and SF-36.

   The Health Assessment Questionnaire (HAQ) is a tool to measure specific functional disability for rheumatoid arthritis. The evaluation covers 8 areas of daily activity. Four types of answers are possible: a score of 0 to 3, where "0" means the absence of disability, while a score of "3" corresponds to a maximum disability.

   The Short Questionnaire to Assess Helath Enhancing Physical Activity (SQUASH) is a questionnaire that assesses average energy expenditure over a week. The questions are grouped into four different themes: commuting activities (going back and forth between home and work / study), leisure activities, home activities, work activity. For each type of activity, it is therefore required to indicate the average time spent per day, the number of days per week and the intensity of effort felt among three possible choices (calm, moderate and intense). The set of reported activities is calculated by multiplying the average time (in minutes) for an activity by its intensity coefficient corresponding to MET intervals. All activity scores are then summed to give the total score.

   The short-form 36 (SF-36) will be used to assess the quality of life and well-being. The SF-36 consists of 36 items, 35 of which are grouped into 8 multi-item scales that measure physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role and mental health. The 8 SF-36 scales are scored on a scale of 0-100, with higher scores indicating a better quality of life.

   During the first session (S1), the target intensity is controlled by monitoring the heart rate as described above. The wattage and pedaling frequency achieved during the first session (S1) will be reproduced for the other series of measurements (S9 and S17).

   The measurements will be carried out at the first session of the protocol (S1) and then every 3 rehabilitation sessions (S5, S9, S13 and S17). These sessions will have a total duration of approximately 75 minutes.
   * (Before exercise) rest extended by 15 minutes; a first evaluation (arterial pressures, elasticity of large and small arteries and the velocity of the radial and distal pulse wave, cutaneous temperature, etc.) of about 7 minutes in the extended position.
   * (After the exercise) second elongated evaluation identical to the previous evaluation. The time between the end of the exercise and the start of the measurement will be controlled and identical for all subjects and measurement series.
   * (After immersion) Third evaluation in lying position identical to the previous evaluation. The time between the end of the immersion and the start of the measurement will be controlled and identical for all subjects and measurements.

   The measurements:
4. / Assessment of arterial stiffness will be performed by analyzing the pressure wave (a) and measuring the velocity of the pulse wave (b).

   a / HDI Pulse WaveTM CR-2000 tonometry device (HDI Hyperdiagnostics Inc., Eagan, Minnesota, USA): measurement of brachial arterial pressures and assessment of compliance of large and small arteries. This device records the shape of the pulse wave at the level of the radial artery using a sensor placed on the wrist (non-invasive measurement): the analysis of the shape of this wave makes it possible to obtain information on the compliance blood. The sensor will be positioned at the radial site used for VOP measurement.

   The HDI device includes a brachial cuff that makes it possible to measure arterial pressures simultaneously with the measurement of arterial stiffness. The systolic and diastolic blood pressure values will be collected at each resting phase.

   b / The assessment of central arterial stiffness will be performed by measuring the pulse wave velocity on the carotid-femoral segment. The evaluation of the arterial stiffness of the territories concerned (legs) or not (arms) by the exercises, will be carried out by the respective measurements of the pulse wave velocity on the carotid-distal and carotid-radial segments. These evaluations are carried out using the complior system (Complior SP®, Artech Medical, Pantin, France).
5. / The skin temperature at the level of the thigh and the arm using a probe for recording the skin temperature: probes MLT409 / A Skin Temperature Probe (transducer ML309 Thermistor Pod - ADInstruments ) fixed on the skin by a hypoallergenic adhesive.
6. / At the end of each exercise, the subject is called to refer to the perception scale Borg, 1998: it goes from 6 to 20 points (where 6 means: "No effort" and 20: "maximum effort" ), and to indicate to the operator the number that corresponds best to the perception of his effort. The Borg Scale provides information on the subject's subjective perception of different parameters, such as stress or pain.
7. / The perception of cold water tolerance will be evaluated with the aid of a visual analogue scale (0-100 mm), at the first, fifth, tenth and fifteenth minute of submerged recovery.

The patient can stop his participation at any time without justification and can ask all the information he wants to the investigator or the operator. In case of exacerbation of the disease in relation to the results of the DAS-28 scale, the patient will leave the study.

The study may be stopped by decision of the competent administrative authority, the sponsor, the coordinating investigator.

Each patient will be able to leave the study by decision of one of these parties but also by decision of a co-investigator or by decision of the interested person himself, according to the regulation and as it is mentioned in the consent .

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) between the ages of 20 and 80, diagnosed with rheumatoid arthritis without any other risk factor in relation to RA, and having a DAS-28 score between 2.6 and 6.
* Signature of informed consent
* Affiliation to a French social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Unstabilized corticosteroids and / or> 10 mg prednisone / day;
* Unstabilized hypertension;
* Pregnant women;
* Alteration of higher functions making comprehension and adherence to a conditioning program impossible (mini mental test <24); Patient who has performed intense physical exercise / physiotherapy within the previous 24 hours the interventions planned in this project;
* Contraindication to immersion in cold water (a dermatological factor and / or vascular or respiratory cardiac dysfunction and / or cold intolerance syndrome and / or syndrome such as Raynaud's Syndrome);
* Inability to perform physical exercise, regardless of its origin (neurological, central or peripheral, cardiovascular or respiratory or musculoskeletal);
* Legal incapacity or limited legal capacity;
* Subject unlikely to cooperate with the study and / or weak cooperation anticipated by the investigator;
* Subject without health insurance;
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File".

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Pressure wave analysis | Week 6
  The tonometry device measures brachial arterial pressures and assessment of compliance of large and small arteries.
  This device records the shape of the pulse wave at the level of the radial artery using a sensor placed on the wrist (non-invasive measurement): the analysis of the shape of this wave makes it possible to obtain information on the compliance blood.
  The device includes a brachial cuff that makes it possible to measure arterial pressures simultaneously with the measurement of arterial stiffness. The systolic and diastolic blood pressure values will be collected at each resting phase.
  This pressure wave analysis will be analysed concomitantly with assessment of central arterial compliance (pulse wave velocity measurement) as a composite outcome of the assessment of arterial compliance in patients following the rehabilitation protocol .
Assessment of central arterial compliance | Week 6
  The assessment of central arterial compliance will be performed by measuring the pulse wave velocity on the carotid-femoral segment.
  The evaluation of the arterial compliance of the territories concerned (legs) or not (arms) by the exercises, will be carried out by the respective measurements of the pulse wave velocity on the carotid-pedal and carotid-radial segments.
  This assessment of central arterial compliance (pulse wave velocity measurement) will be analysed concomitantly with pressure wave analysis as a composite outcome of the assessment of arterial compliance.

SECONDARY OUTCOMES:
Disease activity Score 28 | Week 6
  the rating of pain in joint pressure and joint swelling on the proximal interphalangeal (PPI), metacarpophalangeal (MCP) joints of the hands, wrists, elbows, shoulders and knees.
  This scale will be analysed concomitantly with measurement of certain blood markers of inflammation and an articular ultrasound as a composite outcome of the disease activity.
Disease activity : blood markers of inflammation | Week 6
  Measurement of certain blood markers of inflammation (IL6; PCR; TNF-α) : 3 blood samples of approximately 20 mL of blood will be taken for the subjects who are doing the whole program and only two blood tests for the other subjects. Venous blood samples will be used to determine serum marker concentrations of C-reactive protein inflammation. The assay of two other blood markers of IL-6 inflammation and TNF-α conventionally used in the clinical follow-up of this type of patient will also be performed.
  This measurement of certain blood markers of inflammation will be analysed concomitantly with DAS-28 clinical test and an articular ultrasound as a composite outcome of the disease activity.
Disease activity : articular ultrasound | Week 6
  The articular ultrasound will be performed on 32 joints of the hands, wrists and feet using a qualitative synovitic score in B mode and Doppler mode each rated from 0 to 32, a total score ranging from 0 to 64.
  This articular ultrasound will be analysed concomitantly with DAS-28 clinical test and measurement of certain blood markers of inflammation as a composite outcome of the disease activity.
Cardiovascular function : blood pressure | Week 6
  blood pressure will be assessed before and after the rehabilitation protocol.
  This blood pressure assessment will be analysed concomitantly with heart rate, cardiac index and elasticity of large and small arteries as a composite outcome of cardiovascular function.
Cardiovascular function : cardiac index | Week 6
  The cardiac index will be assessed before and after the rehabilitation protocol.
  The cardiac index corresponds to the quotient of the left ventricular cardiac output per minute by the body surface, thus connecting the cardiac performance to the size of the individual. The unit of measure is liter per minute per square meter (L / min / m2).
  This cardiac index assessment will be analysed concomitantly with blood pressure assessment, heart rate and elasticity of large and small arteries as a composite outcome of cardiovascular function.
Cardiovascular function : elasticity of arteries | Week 6
  The elasticity of large and small arteries will be assessed before and after the rehabilitation protocol.
  This elasticity of arteries assessment will be analysed concomitantly with blood pressure assessment, heart rate and cardiac index as a composite outcome of cardiovascular function.
Assessment of functional disability : HAQ | Week 6
  The Health Assessment Questionnaire (HAQ) is a tool to measure specific functional disability for rheumatoid arthritis.
Assessment of physical activity (SQUASH) | Week 6
  The Short Questionnaire to Assess Helath enhancing physical activity (SQUASH) is a questionnaire to evaluate the average energy expenditure during a week.
Assessment of quality of life and well-being (SF-36) | Week 6
  The Short-forme 36 (SF-36) questionnaire will be used to assess the quality of life and well-being.
  This SF-36 questionnaire will be analysed concomitantly with HAQ and SQUASH questionnaires as a composite outcome of the assessment of functional disability, physical activity and quality of life and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Clément Prati, Besançon, France